CLINICAL TRIAL: NCT05698290
Title: Engaging School Providers to Manage Student Pain in Michigan Schools
Brief Title: HELP Pain Training Program
Status: Active, not recruiting | Type: Observational
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Natoshia Cunningham, Assistant Professor, Michigan State University
Other Study IDs: STUDY00007400
Record Dates: First submitted 2022-11-29; First posted 2023-01-26 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pain
Keywords: Pain; Cognitive Behavioral Therapy; School Providers
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health Department of Northwest Michigan: School providers (school nurses, mental health specialists) from the Health Department of Northwest Michigan.
  Interventions: Other: HELP Pain Training Program
- Michigan Association of School Nurses: School providers (nurses) from the Michigan Association of School Nurses.
  Interventions: Other: HELP Pain Training Program

INTERVENTIONS:
Other: HELP Pain Training Program — A training program to teach school providers nonpharmacologic (e.g., cognitive behavioral and mindfulness meditation) strategies to use with students with pain symptoms.

SUMMARY:
The aim of this project is to develop and test the Helping Educators Learn Pediatric Pain Assessment & Intervention Needs (HELP Pain) program. HELP Pain provides training for school providers (e.g., school nurses, mental health professionals) on strategies to assess and manage pain-related concerns in school children. Participants will learn cognitive behavioral therapy techniques to help school children manage pain, and report on their use of strategies, and child's progress throughout the school year. Follow-up data will be collected in year 2.

DETAILED DESCRIPTION:
Chronic pain is common among school children, and impacts social, emotional and academic functioning. School providers are often tasked with addressing student pain, but may have limited training in evidence-based pain management strategies. Thus, the PI developed a training program, HELP Pain, to train school providers, such as school nurses and mental health professionals, in cognitive behavioral therapy strategies for addressing student pain. In this study, the feasibility and acceptability of the training program will be evaluated. Provider knowledge will be evaluated before and after receiving the HELP Pain training. Further, the use of HELP Pain strategies with students and their associated disability and pain outcomes will be evaluated. Results will help to tailor the HELP Pain training program for future use.

ELIGIBILITY:
Inclusion Criteria:

* engaged as a school provider in Michigan

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Providers (nurses and mental health professionals) serving Michigan schools.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Qualitative report | 9 months
  Implementation success of the program measured by a semi-structured qualitative interview method which addresses feasibility.
Acceptability - Qualitative report | 9 months
  Implementation success of the program measured by a semi-structured qualitative interview method which addresses acceptability.
Appropriateness - Qualitative report | 9 months
  Implementation success of the program measured by a semi-structured qualitative interview method which addresses appropriateness.
Implementation Success - Quantitative report | 9 months
  Twelve psychometrically validated items to assess program implementation success, will be administered after training. Providers will rate items with responses using a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5).

SECONDARY OUTCOMES:
Knowledge | 9 months
  Knowledge quiz scores before and after training, 0-20, where 20 indicates higher knowledge.
Fidelity | 9 months, 2 years
  Self-reported use of HELP Pain strategies with students via online survey.
Self-report Knowledge | 9 months
  Self-reported agreeableness using a 5-point Likert scale from strongly disagree (1) to strongly agree (5) to 3 statements indicating knowledge from the program.

OTHER OUTCOMES:
Child Functional Disability Inventory (FDI) | 9 months, 2 years
  Administration of the FDI to students is optional. The FDI is used to assess impairment due to pain over the past several days, and uses a Likert scale (0-4) to result in a score 0-60, where 60 implies decreased functioning.
Child Pain Ratings - Numerical Scale | 9 months, 2 years
  Administration of the child pain ratings to students is optional. Highest, lowest, average and current pain over the past week are reported by a child to the provider using a numerical scale. The numerical scale is 0-10, with 10 indicating worse pain.
Child Pain Ratings - Faces Scale | 9 months, 2 years
  Administration of the child pain ratings to students is optional. Highest, lowest, average and current pain over the past week are reported by a child to the provider using a faces scale. The faces scale contains 6 faces with scores of 0, 2, 4, 6, 8, or 10 respectively from left to right, where the rightmost face or score of 10 indicates worse pain.
Child School Attendance | 9 months, 2 years
  Reporting of a child's school attendance is optional. School attendance, late arrivals, and early dismissal in one month (due to pain or other reasons), and school nurse visits for pain or other reasons (scheduled and unscheduled) as reported by the school provider specific to a child.

CONTACTS AND LOCATIONS:
Overall Officials: Natoshia R Cunningham, Ph.D., Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, Grand Rapids, Michigan, United States